CLINICAL TRIAL: NCT00677950
Title: OP-1 Putty for Posterolateral Fusions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olympus Biotech Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S01-01US
Record Dates: First submitted 2008-05-13; First posted 2008-05-15 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Degenerative Lumbar Spondylolisthesis
Keywords: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — Spinal Fusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): OP-1 Putty
  Interventions: Procedure: Spinal fusion
- 2 (Active Comparator): Autograft
  Interventions: Procedure: Spinal fusion

INTERVENTIONS:
Procedure: Spinal fusion — Surgical procedure for lumbar spinal posterior decompression with concomitant posterolateral intertransverse process arthrodesis
  Other Names: Lumbar Spinal Fusion

SUMMARY:
The trial was designed to demonstrate the comparability of the overall success rate in the OP-1 Putty treatment group to the autograft treatment group.

DETAILED DESCRIPTION:
A controlled, open- label, blinded radiographic assessment, randomized, prospective, multicenter, multinational pivotal study in which patients with single level (L3-S1) degenerative lumbar spondylolisthesis (Grade 1 or 2) with spinal stenosis underwent decompression and spinal fusion and received OP-1 Putty or autograft. This study was a one-sided, non- inferiority trial comparing the overall success between the OP-1 Putty group and the control autograft group.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has a diagnosis of Degenerative Lumbar Spondylolisthesis of Grade I or II with Spinal Stenosis demonstrated by medical history, physical examination a n d radiographic imaging.
2. The subject is a candidate for decompression and spinal fusion with the use of autograft from the iliac crest.
3. The subject requires one level lumbar fusion (L-3 to S-1).
4. The subject has a preoperative Oswestry Disability Index of 30-100.

Exclusion Criteria:

1. The subject has active spinal and/or systemic infection.
2. The subject is morbidly obese.
3. The subject has a known sensitivity to any component of the OP-1 Putty.
4. The subject has spinal instability measured on flexion / extension radiographs of greater than 50% translation of the vertebrae and greater than or equal to 20 degrees of angular motion.
5. The subject uses tobacco or nicotine or is prescribed steroids such as cortisone.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2001-10; Primary Completion 2003-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Overall success rate at 24 months in the OP-1 Putty and the autograft groups, radiographic demonstration of spinal fusion, ODI improvement of at least 20%, no revisions, removals or supplemental fixations | 3, 6, 12, 24 months

SECONDARY OUTCOMES:
The number of anticipated and unanticipated complications/AEs that occurred within the study population, Visual Analog Scale Results for Pain Assessment, Donor Site Pain, Medication Use | 3, 6, 12, 24 months

CONTACTS AND LOCATIONS:
Locations (24):
- United States (21):
  - Santa Monica, California
  - Stanford, California
  - Denver, Colorado
  - Newark, Delaware
  - Clearwater, Florida
  - Fort Lauderdale, Florida
  - Miami, Florida
  - Chicago, Illinois
  - Kalamazoo, Michigan
  - Southfield, Michigan
  - St Louis, Missouri
  - New York, New York
  - Rochester, New York
  - Charlotte, North Carolina
  - Akron, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Germantown, Tennessee
  - San Antonio, Texas
  - Charlottesville, Virginia
  - Fairfax, Virginia
- Canada (3):
  - Halifax, Nova Scotia
  - London, Ontario
  - Toronto, Ontario